CLINICAL TRIAL: NCT05942534
Title: Pediatric Mask Fit Study: Comparing the Performance of Cloth Masks, Procedure Masks With and Without Modifications and Respirators in Children
Brief Title: Pediatric Mask Fit Study
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michelle Science, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000080453
Record Dates: First submitted 2023-06-16; First posted 2023-07-12 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mask type assessment: The mask type assessment will compare a cloth mask, child and adult medical mask, child and adult KN95 respirator, and N95 respirator.
- mask modification assessment: The mask modification assessment will compare a child medical mask, adult medical mask with and without modifications (tuck and tie, twisted ear loops), and child and adult N95 respirator.

SUMMARY:
This study will evaluate the performance of various face masks and respirators on children by examining their fitted filtration efficiency (FFE) and mask fit. It will also evaluate the impact of different types of mask modifications (for example, twisting the ear loops, tuck and tie) on FFE and mask fit, with the goal of determining how to optimize mask performance in children. It will also provide information on mask and respirator comfort and acceptability. This data will help inform public health messaging around mask choice for children and also modifications that can be made to improve fit for children who may not have access to various mask types.

DETAILED DESCRIPTION:
This will be a prospective cross-sectional study of 200 children aged 4 to 17 years. Participants will be assigned to either the mask type assessment (Objective 1) or the mask modification assessment (Objective 2) and have a date and time scheduled for testing.

The mask type assessment will compare the FFE and fit factor of a cloth mask, child and adult medical mask, child and adult KN95 respirator, and N95 respirator. The mask modification assessment will compare the FFE and fit factor of a child medical mask, adult medical mask with and without modifications (tuck and tie, twisted ear loops), and child and adult N95 respirator. Quantitative fit testing will be conducted using a TSI Portacount Pro Respirator Fit Tester model 8038+. Testing will be performed in an identified designated area at the hospital or in the community (i.e., schools or community center), monitored for ventilation, temperature and humidity. We will also measure the ambient particles to ensure adequate particle count. The participants will be asked to evaluate the mask, respirator or modification based on a variety of criteria including comfort, breathability and acceptability. This will be completed immediately after the fit assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 4-17
* able to tolerate wearing a mask

Exclusion Criteria:

* Children will be excluded if they have contraindications to wearing a mask.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 4 to 17 years able to wear a mask
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-29 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Fitter filtration efficiency and fit factor | First visit (1 hour)
  To compare the performance of different mask (cloth and medical) and respirator (KN95 and N95) types and mask modifications in children, as measured by fitted filtration efficiency (FFE) and fit factor.

SECONDARY OUTCOMES:
Mask and respirator comfort and acceptability | First visit (1 hour)
  Evaluate the comfort and acceptability of different masks, mask modifications, and respirators as experienced by children

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No